CLINICAL TRIAL: NCT00371969
Title: Reducing Unsafe Drinking in HIV Primary Care
Brief Title: Reducing Unsafe Alcohol Use in HIV-Positive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Deborah Hasin, Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-HAS-14323; NIH Grant R01 AA14323-01A1
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Alcohol Abuse
Keywords: Unsafe drinking; Human Immunodeficiency Virus; Motivational Interviewing
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome

ARMS (2):
- 1 - enhanced MI (Active Comparator): Enhanced brief motivational interview (including an IVR component for alcohol self-monitoring purposes)
  Interventions: Behavioral: Enhanced Motivational Interview
- 2- standard MI (Active Comparator): The intervention consists of a standard motivational interview or viewing a DVD on HIV self-care.
  Interventions: Behavioral: Standard Motivational Interview or viewing DVD

INTERVENTIONS:
Behavioral: Enhanced Motivational Interview — The intervention consists of a brief motivational interview, which is combined with daily alcohol monitoring through the use of an interactive voice response system IVR (automated telephone system).
  Arms: 1 - enhanced MI
Behavioral: Standard Motivational Interview or viewing DVD — Brief motivational interview, viewing a DVD on HIV self-care.
  Arms: 2- standard MI

SUMMARY:
The main aim of this study is to test an intervention to reduce unsafe drinking among HIV-positive primary care patients. The intervention consists of a brief motivational interview, which is combined with daily alcohol monitoring through the use of an interactive voice response system IVR (automated telephone system). Subjects who receive the enhanced motivational interview are expected to show greater improvements in drinking than individuals who receive the standard motivational interview or view a DVD on HIV self-care.

DETAILED DESCRIPTION:
HIV infection is a widespread health problem in the U.S. Antiretroviral treatment has increased longevity and changed the nature of risk factors for morbidity and mortality. Alcohol consumption has become an increasingly serious health issue among HIV primary care patients. Drinking is a key factor in progression to severe liver damage (especially those co-infected with hepatitis), and liver disease is now one of the most common causes of death among those with HIV. Excess drinking is also associated with medication noncompliance, reduces the effect of antiretroviral treatment, and is linked to other health problems. Therefore, helping HIV patients reduce unsafe drinking is crucial to their long-term health. The intervention combines the brief MI, an established, evidence-based counseling approach, with an innovative procedure designed to strengthen the effects of the MI. An effective, easily implemented alcohol-reduction intervention could be incorporated into standard care in HIV clinics helping prevent or slow the progress of some medical problems in HIV-infected individuals, improve medication compliance, prolong lifespan and decrease risk behavior associated with alcohol use.

Comparison(s): Enhanced brief motivational interview (including an IVR component for alcohol self-monitoring purposes), brief motivational interview, viewing a DVD on HIV self-care.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older.
* Participants have had 4 or more drinks on any day in the prior 30 days assessed via standardized questions.
* Participants are referred to a study MI counselor by clinic staff as needing an intervention for drinking
* Participants agree to random assignment and provide informed consent

Exclusion Criteria:

* Participants who are currently psychotic, suicidal or homicidal.
* Participants who have definite plans to leave the greater New York metropolitan area within the study period.
* Participants who demonstrate gross cognitive impairment as evidenced on the Halstead-Reitain Trails (A).
* Participants who do not speak English or Spanish, or have hearing impairments that preclude use of the telephone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption in the last 30 days, assessed at baseline and repeatedly during follow-up so that change can be analyzed. | Baseline, 30, 60 days (end-of-treatment), 3, 6, 12 months
  As measured by number of drinks per drinking day and percentage of days abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Selvija G. Marovic, PhD, Study Director — New York State Psychiatric Institute (NYSPI)
Locations (1):
- New York State Psychiatric Institute/ St. Vincent's Hospital, New York, New York, United States

REFERENCES:
- [Derived] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593